CLINICAL TRIAL: NCT02451319
Title: Comparison of Safety and Efficiency of 20w 30w Holmium Laser Device in Treatment of 1-2 cm Diameter Kidney Stones With RIRS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Nihat Karakoyunlu, MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 26.01.2015 19/17
Record Dates: First submitted 2015-04-28; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Nephrolithiasis
Keywords: RIRS, holmium, 1-2 cm,stones,kidney
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- first group (Active Comparator): Patients undergoing Retrograde Intrarenal Surgery with 20w holmium laser device who have 1-2 cm diameter kidney stones
  Interventions: Procedure: Retrograde Intrarenal Surgery
- second group (Active Comparator): Patients undergoing Retrograde Intrarenal Surgery with 30w holmium laser device (working over 20w power) who have 1-2 cm diameter kidney stones
  Interventions: Procedure: Retrograde Intrarenal Surgery
- third group (Active Comparator): Patients undergoing Retrograde Intrarenal Surgery with 30w holmium laser(working under 20w power) device who have 1-2 cm diameter kidney stones
  Interventions: Procedure: Retrograde Intrarenal Surgery

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery — Endoscopic treatment of Kidney Stones

SUMMARY:
To compare the safety and Efficiency of 20w 30w holmium laser device in treatment of 1-2 cm diameter kidney stones with Retrograde Intrarenal Surgery (RIRS).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 18-90 years old
* Patients undergoing RIRS for treatment of 1-2 cm diameter kidney stones

Exclusion Criteria:

* Patients who have congenital urogenital abnormalities
* Patients who have previous stone surgery history

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Safety - complications according to clavien system | postoperative 24 hours
  complications according to clavien system
safety - visual analog score | postoperative 24 hours
  visual analog score

SECONDARY OUTCOMES:
efficiency - stone free rate | postoperative 24 hours
  stone free rate post operative first day

CONTACTS AND LOCATIONS:
Overall Officials: Nihat Karakoyunlu, MD, Principal Investigator — Dıskapı TRH
Locations (1):
- Tuekey Ministry of HealthDıskapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Redondo C, Ramon de Fata F, Gimbernat H, Meilan E, Andres G, Angulo JC. Retrograde intrarenal surgery with holmium-YAG laser lithotripsy in the primary treatment of renal lithiasis. Actas Urol Esp. 2015 Jun;39(5):320-6. doi: 10.1016/j.acuro.2014.06.004. Epub 2014 Oct 25. English, Spanish. PMID 25443519